CLINICAL TRIAL: NCT01717664
Title: A Phase IIa Proof of Concept Study to Assess the Efficacy and Safety of Fixed Dose Combination RHB-104 as Add-On Therapy to Interferon Beta-1a in Patients Treated for Relapsing Remitting Multiple Sclerosis
Brief Title: Proof of Concept Study of RHB-104 as Add-On Therapy to Interferon Beta-1a in Relapsing Remitting Multiple Sclerosis (RRMS)
Acronym: CEASE-MS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHB-104-02
Record Dates: First submitted 2012-10-24; First posted 2012-10-30 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis; MAP; antibiotic; Interferon beta 1-a; MS; MRI; EDSS; relapse rate
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RHB-104 (Experimental): 5 RHB-104 capsules administered orally BID
  Interventions: Drug: RHB-104

INTERVENTIONS:
Drug: RHB-104 — 95 mg clarithromycin, 45 mg rifabutin, and 10 mg clofazimine

SUMMARY:
The investigators hypothesize that Mycobacterium avium paratuberculosis positive Relapsing Remitting MS subjects will have a greater response to Interferon beta-1a therapy plus RHB-104 than from Interferon beta-1a alone.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥18 years
* Signed fully informed consent provided as per this protocol and willing to comply with the required scheduled assessments of the protocol.
* Diagnosis of relapsing-remitting multiple sclerosis (McDonald Criteria (2010)) with dissemination in time and space.
* Currently treated with a stable dose of Rebif®, or Avonex® for a minimum of 3 months duration prior to the screening visit.
* Active MS with history of at least one flare within the past 12 months or two flares in the past 24 months prior to screening.
* An Expanded Disability Status Scale (EDSS) of 6.0 or less at the screening visit.
* White blood cell count ≥ to 3.5x109.
* Subject agrees to use barrier contraceptive methods (i.e. diaphragm, cervical cap, contraceptive sponge or condom) with spermicidal foam/gel/cream/suppository, or IUD from study enrolment through 6 weeks after last dose of study medication, unless subject is post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation, or has had a vasectomy. Subject agrees to appropriate contraception method though completion of study.

Exclusion Criteria:

* Treatment with any other biological therapies including but not limited to Interferon beta-1b, natalizumab, anti-TNF biologic agents, or other agents intended to reduce TNF ≤ 8 weeks prior to screening or within 5 half-lives of agent prior to screening, whichever is longer.
* Previous treatment with rifabutin and/or clofazimine.
* Previous treatment with amiodarone.
* Oral or parenteral antibiotics in the 4 weeks prior to screening. (Topical antibiotics are permitted.)
* Use of Methylprednisolone sodium succinate, prednisone, or any other corticosteroid during the 30 days prior to screening.
* Relapse within the 30 days prior to screening, or between screening and baseline.
* Initiation or dose modification of 4-aminopyridine within 60 days of screening.
* Use of azathioprine, 6-mercaptopurine (6-MP), methotrexate, cyclosporine or mycophenolate (CellCept) within 8 weeks prior to screening.
* Use of glatiramer acetate, cyclophosphamide, or plasma exchange within 12 weeks prior to screening.
* Use of mitoxantrone within one year prior to screening.
* Any previous treatment with cladribine, T cell vaccine, or altered peptide ligand.
* Previous total body irradiation or total lymphoid irradiation.
* Treatment with any medication that causes QT prolongation or Torsades de Pointes within 7 days prior to initiation of study drug, including but not limited to: Cisapride, pimozide, astemizole, terfenadine, ergotamine, dihydroergotamine, quinidine, procainamide, disopyramide, sotalol, ibutilde, dofetilide, dronedarone, ondansetron or other 5-HT3 receptor agonists, citalopram dose greater than 20 mg/day, tolteridine and quinine.
* Treatment with the following medications within 7 days prior to initiation of study drug: colchicine, roflumilast, apixabin, latuda, nefazodone, buspirone, fluvoxamine, simvastatin, lovastatin, atorvastatin, amlodipine, diltiazem, felodipine, nifedipine, nitrendipine, nisoldipine, fluconazole, ketoconazole, voriconazole, St. Johns wort, grapefruit juice, antiretroviral agents, alprazolam, alfentanyl, aprepitant, aripiprazole, cyclosporine, boceprevir, carbamazepine, haloperidol, digoxin, propranolol, carvedilol, metoprolol, and estrogens.
* Adverse reaction or hypersensitivity to the study drug or any medications related to the study drug.
* Clinically significant abnormalities of hematology or chemistry at screening as confirmed by repeat testing based on investigator's discretion, including but not limited to, elevations greater than 2 times the upper limit of normal of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), or creatinine clearance less than 60 ml/min at screening.
* Serum potassium, magnesium or calcium outside the normal reference range considered clinically significant by the investigator.
* Positive stool results for C. difficile.
* A positive serology for Hepatitis B, Hepatitis C or HIV at screening except for the following:

If positive history of previously treated Hepatitis C, but HCV PCR is undetectable off medications for at least 6 months prior to screening, and treating hepatologist or infectious disease specialist believes the subject is cured - subject may be enrolled

* One of the following:

History of atypical mycobacterial infections (other than MAP). History of active tuberculosis (TB) requiring treatment in the past 3 years. Tuberculosis infection as determined by a positive diagnostic TB test result (defined as a positive or indeterminate (after two independent tests) quantiFERON TB Test Gold test).

* Currently diagnosed or history of uveitis confirmed by either an ophthalmologist or optometrist.
* Any evidence of any other significant hematological, hepatic, renal, cardiac, pulmonary, metabolic, thyroid, neurological or psychiatric disease that might interfere with the subject's ability to safely enter and or complete the study requirements.
* History of malignancy within the past five years except for basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
* Males who do not use barrier contraceptive methods (i.e. condom) with spermicidal foam/gel/cream/suppository or have not had a vasectomy.
* Females who:

  1. have a positive pregnancy test
  2. are lactating
* Refusal to sign the study informed consent form.
* Inability to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study.
* History of drug or alcohol abuse within the past 3 years.
* Participation in any experimental drug protocol within 12 weeks of date of screening.
* Cardiac pacemaker or any other type of metal implant or any other contraindication for MRI (including known allergy to gadolinium).
* QTc greater than 440ms, bundle branch block, or major ST or T wave abnormalities that make the assessment of the QT impossible.
* History of unstable cardiac syndromes including unstable angina, coronary artery bypass graft, myocardial infarction or coronary stenting within 2 months of screening; NYHA Class 3-4 CHF; history of ventricular tachycardia, ventricular fibrillation, personal or family history of sudden death, Long QT Syndrome, or Torsade de Pointes; HR<50BPM; having taken any Class 1 or Class 3 antiarrhythmic medications or medicines known to prolong the QT interval or be associated with Torsade de Pointes.
* Treatment with medical cannabis in the 4 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Combined Unique Active lesions | Baseline through Wk 24

OTHER OUTCOMES:
Combined Unique Active lesions | Week 24 to Week 48
Change in cytokine panel | Baseline to Week 24
Change in cytokine panel | Week 24 to Week 48
MAP status as established by polymerase chain reaction (PCR) | Baseline to Week 24
MAP status as established by polymerase chain reaction (PCR) | Week 24 to Week 48
Relapses | Baseline to Week 24
Relapses | Week 24 to Week 48
Expanded Disability Status Scale (EDSS) | Baseline to Week 24
Expanded Disability Status Scale (EDSS) | Week 24 to Week 48
T2-hyperintense lesions | Baseline to Week 24
T2-hyperintense lesions | Week 24 to Week 48
T1 post-gadolinium lesions | Baseline to Week 24
T1 post-gadolinium lesions | Week 24 to Week 48
Burden of Disease | Baseline to Week 24
Burden of Disease | Week 24 to Week 48
Number of participants with adverse events | Baseline through Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Ira N Kalfus, MD, Study Director — RedHill Biopharma; Radi Shahien, MD, Principal Investigator — Ziv Medical Center
Locations (2):
- Israel (2):
  - RedHill MS Clinical Trial Site 002, Tel Aviv
  - RedHill MS Clinical Trials Site 001, Zefat (Safed)